CLINICAL TRIAL: NCT04991038
Title: Prospective, Multi-center, Randomized Study to Compare the Safety and Efficacy of the DAISe Thrombectomy System and Stent Retrievers for Neurointervention in Acute Ischemic Stroke
Brief Title: Clinical Investigation to Compare Safety and Efficacy of DAISE and Stent Retrievers for Thrombectomy In Acute Ischemic Stroke Patients
Acronym: DAISE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn, considering alternative trial design
Sponsor: MIVI Neuroscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 101903
Record Dates: First submitted 2021-07-27; First posted 2021-08-05 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Stroke; Stroke, Ischemic; Stroke, Acute; Cerebrovascular Disorders; Cerebrovascular Accident
Keywords: DAISE; thrombectomy
MeSH Terms: conditions — Stroke; Ischemic Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- DAISe Thrombectomy Device (Experimental): Mechanical Thrombectomy with DAISe
  Interventions: Device: DAISe Device
- Stent Retriever (Active Comparator): Mechanical Thrombectomy with TREVO or Solitaire Device
  Interventions: Device: Trevo or Solitaire

INTERVENTIONS:
Device: DAISe Device — Thrombectomy using the DAISE device
  Arms: DAISe Thrombectomy Device
Device: Trevo or Solitaire — Thrombectomy using TREVO or Solitaire device
  Arms: Stent Retriever

SUMMARY:
Compare the safety and efficacy of the DAISE to stent retrievers in the treatment of acute ischemic stroke

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Pre-stroke independent functional status in activities of daily living with modified Rankin Score 0-1
* Patient presenting with a disabling stroke device as NIHSS ≥6
* Thrombolytic therapy (IV tPA), if indicated/administered, was initiated within 3 hours of onset/ last known well according to prescribed dosing.Endovascular treatment intended to be initiated (groin puncture) <24 hours from onset of symptoms or last known well time.
* Confirmed symptomatic large vessel occlusion of the intracranial internal carotid artery, M1 or proximal M2 segment of the middle cerebral artery.
* The following image criteria should also be met:

For Subjects 0-6hrs onset:

* MRI Criterion: volume of diffusion restriction as assessed by automated core volume software ≤50mL OR
* CT Criterion: ASPECTS 6-10 on baseline CT or CTA-source images or, CPT as assessed by automated core volume software ≤50mL

For subjects 6-24hrs onset:

* ≤20mL Ischemic core volume if age >80
* ≤30mL Ischemic core volume if age <80 and NIHSS 10-20
* ≤50mL Ischemic core volume if age <80 and NIHSS >20
* Signed informed consent from patient or legal authorized representative.

Exclusion Criteria:

* CT or MRI evidence of intracranial hemorrhage on presentation.
* CT or MRI showing mass effect or intracranial tumor (meningioma >2cm in diameter)
* CT or MRI evidence of carotid dissection or complete cervical carotid occlusion requiring a stent.
* Previous stroke within the past 3 months.
* Known arterial condition (proximal vessel stenosis or pre-existing stent) that would prevent the study devices from reaching the target vessel and/or preclude safe recovery of the study devices.
* Pregnancy.
* Severe contrast allergy or absolute contraindication to iodinated contrast.
* Rapidly improving neurological status as determined by Investigator/Neurologist.
* Renal failure/insufficiency with >3.0 mg/dL creatinine prior to procedure.
* Severe, sustained hypertension resistant to treatment (SBP>185mmHg or DBP >110mmHg)
* Use of warfarin anticoagulation with International Normalized Ratio (INR) >3.0 at the time of the procedure or any known hemorrhagic or coagulation deficiency.
* For patients who have received a direct thrombin inhibitor within the last 48hrs; partial thromboplastin time (PTT) > 2.0 times the normal prior to procedure.
* Platelet count < 50,000
* Cerebral vasculitis or evidence of active systemic infection (including COVID-19)
* Suspicion of aortic dissection, septic embolus, or bacterial endocarditis.
* Clinical symptoms suggestive of bilateral stroke or occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation).
* Seizure due to stroke.
* Clinical history, past imaging or clinical judgment suggests that the intracranial occlusion is chronic.
* Active participation in another study involving an investigational drug or device.
* A severe or fatal comorbid illness that will prevent improvement or follow-up or that will render the procedure unlikely to benefit the patient.
* Unwillingness to complete follow up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Outcome: Good Functional Outcome of Modified Rankin Score 0-2 | 90 days
Primary Safety Outcome: Symptomatic intracranial hemorrhage | 24hrs post procedure

SECONDARY OUTCOMES:
mTICI 2b-3 after randomized modality | procedure after use of randomized device
mTICI 2b-3 after first attempt with randomized modality | procedure after first attempt with randomized device
mTICI 2c-3 after randomized modality | procedure after use of randomized device
mTICI 2c-3 after the first attempt with randomized modality | procedure after first attempt with randomized device
mTICI 2b-3 at end of the procedure | procedure after all interventions
mTICI 2c-3 at end of the procedure | procedure after all interventions
Procedure Time | procedure
  Time from groin puncture to first successful revascularization devices as mTICI 2b-3 flow (as long as final mTICI 2b-3 is achieved)
Rates of procedure and/or device related serious adverse events | 90 days
Rate of all intracranial hemorrhage at 24hrs | 24hrs
Rate of embolization to a new vascular territory (ENT) during procedure | procedure
All-cause mortality at 90 days | 90 days
Neurologic/Stroke related mortality at 90 days | 90 days
Patient reported outcome assessment by PROMIS Global-10 at 90 days | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Siddiqui, MD, PhD, Principal Investigator — UB/Kaleida Health; Brian Jankowitz, MD, Principal Investigator — U Penn Medical Center; Luvas Elijovich, MD, Principal Investigator — University of Tennessee Health Sciences Center

IPD SHARING:
Plan to Share IPD: No